CLINICAL TRIAL: NCT01901159
Title: A Randomized, Single Dose, Open-label, Two Parts, Two and Three Period Cross-over Study to Investigate the Relative Bioavailability of Two Tablet Formulations and the Effect of Fasting Following Oral Administration of RO4995819 in Healthy Subjects
Brief Title: A Study of RO4995819 to Assess Bioavailability and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BP28433; 2012-002710-39 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-07-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- RO4995819 capsule (Experimental)
  Interventions: Drug: RO4995819
- RO4995819 tablet (Experimental)
  Interventions: Drug: RO4995819

INTERVENTIONS:
Drug: RO4995819 — Oral doses of RO4995819 (tablet)
  Arms: RO4995819 tablet
Drug: RO4995819 — Oral doses of RO4995819 (capsule)
  Arms: RO4995819 capsule

SUMMARY:
This randomized, open-label, cross-over study will assess the bioavailability and safety of RO4995819 in healthy volunteers. Volunteers will receive two different formulations (tablet and capsule) of the study drug under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male and female volunteers, 18 to 65 years of age, inclusive.
* A body mass index (BMI) between 18 to 30 kg/m2, inclusive.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.
* Willing not to participate in any other clinical trial with an investigational drug or device for at least 3 months following the follow up visit.
* Male volunteers and their partners of childbearing potential must use two adequate methods of contraception. Female volunteers who are not either surgically sterile or postmenopausal must commit to use two adequate methods of contraception throughout the study and until at least 5 months after last dosing.

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder or cancer
* Significant past or present disorders of the central nervous system, psychiatric disorders, behavioral disturbances
* Diseases or medical conditions that are capable of altering the absorption, metabolism or elimination of drugs
* Any condition or disease detected during the medical interview / physical examination that would render the volunteer unsuitable for the study, place the volunteer at undue risk or interfere with the ability of the volunteer to complete the study in the opinion of the Investigator
* Clinically significant abnormalities in laboratory test results
* Confirmed resting pulse rate greater than 90 or less than 40 beats per minute (bpm) at screening
* Confirmed systolic blood pressure (SBP) greater than 140 or less than 90 mm Hg, and diastolic blood pressure (DBP) greater than 90 or less than 50 mm Hg at screening
* Any major illness within the 4 weeks prior to dosing or any acute disease state within 7 days of study start
* Any confirmed allergic reaction against any drug or multiple allergies
* Any suspicion or history of alcohol abuse and/or consumption of other drugs of abuse
* Infection with hepatitis B, hepatitis C virus, or HIV 1 and HIV 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability: Plasma concentration of RO4995819 | Approximately 3 months

SECONDARY OUTCOMES:
Safety: incidence of adverse events | Approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France